CLINICAL TRIAL: NCT06294470
Title: Efficacy of the Hemorrhoidal Prolapse and Pexia Procedure for the Treatment of Defecatory Obstruction Syndrome.
Brief Title: Efficacy of Stapled Hemorrhoidopexy for the Treatment of Obstructive Defecation Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Central de Venezuela (Other)
Responsible Party: Principal Investigator, Cristopher Varela, M.D., Universidad Central de Venezuela
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-2023
Record Dates: First submitted 2024-01-30; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Hemorrhoids; Defecation Disorder
Keywords: Hemorrohoids; Obstructive Defecation Syndrome; Stapled hemorrhoidopexy
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Altomare Score score ≥3pts and Agachan Wexner Score ≥12pts
  Interventions: Diagnostic Test: Ballon expulsion test; Diagnostic Test: Colonic transit time; Procedure: Stapled hemorrhodopexy
- Control (Active Comparator): Altomare Score score <3pts and Agachan Wexner Score <12pts
  Interventions: Diagnostic Test: Ballon expulsion test; Diagnostic Test: Colonic transit time; Procedure: Stapled hemorrhodopexy

INTERVENTIONS:
Diagnostic Test: Ballon expulsion test — Rectal latex balloon probe filled with saline solution. Patients expelled balloon and time recorded (<1 or >1 min).
Diagnostic Test: Colonic transit time — Patients ingested capsules with 24 radiopaque markers and underwent standing abdominal radiographs on Day 3 and Day 5. Over 80% expulsion within five days was considered normal, while retention indicated defecatory obstruction.
Procedure: Stapled hemorrhodopexy — Circumferential stapled hemorrhoidopexy with a 34mm circular stapler is a surgical procedure used to treat mucohemorrhoidal prolapse.

SUMMARY:
The objective of this study is to assess the efficiency of the procedure for hemorrhoidal prolapse and pexia in alleviating symptoms of defecatory obstruction among patients with grade II to IV mucohemorrhoidal prolapse.

DETAILED DESCRIPTION:
In 1998, Longo introduced a new technique called the stapled hemorrhoidal prolapse and pexia procedure (PPH) to treat mucohemorrhoidal disease. According to Longo, hemorrhoidal prolapse is always associated with internal rectal prolapse, which can be a symptom of defecation obstruction syndrome. The PPH technique aims to correct these symptoms by removing the mucosal segment and pexiing the hemorrhoids, thus eliminating excess rectal tissue. This improves the resting surface tension of the rectal mucosa, making defecation easier and improving defecatory obstruction.

The research focused on applying theoretical concepts related to defecatory obstruction secondary to mucohemorrhoidal prolapse, which results in difficulties with an adequate defecatory act. The main objective was to determine if surgery for hemorrhoidal prolapse and pexia could correct the symptoms of obstructed defecation, as proposed by Longo. The study established facilities to evaluate and provide pre- and postoperative follow-up to patients with symptoms of defecatory obstruction. The research question posed was: "In patients with mucohemorrhoidal disease and symptoms of defecatory obstruction, can the PPH technique improve the symptoms of defecatory obstruction?"

To carry out the research, a questionnaire was used to collect epidemiological, clinical, and functional data from patients with grade II to IV mucohemorrhoidal disease who had surgical indication for PPH. The Constipation Scores questionnaire (Altomare and Agachan-Wexner) was used to identify patients with symptoms of defecatory obstruction. The sample was divided into two groups: an experimental group, which included patients with symptoms of defecatory obstruction, and a control group, made up of patients without such symptoms. Functional studies were carried out, such as colonic transit time and the balloon expulsion test. Subsequently, the PPH technique was performed, and after one month postoperatively, the Constipation Scores and functional studies were evaluated to determine if there was an improvement in the initial scores.

The study was designed as a quasi-experimental study and was also supported by an analytical case-control study. Its aim was to assess patients with grades II to IV mucohemorrhoidal disease who required PPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years old.
* Patients diagnosed with grade II to IV mucohemorrhoidal disease and suffering from symptoms of obstructed defecation, which require a procedure for prolapse and hemorrhoidal pexia.
* Patients with a minimum Altomare Score of 3pts and Agachan Score Wexner of at least 12pts.

Exclusion Criteria:

* Patients who, after undergoing a colonic transit time study, are found to have a different type of constipation (such as slow transit or colonic inertia).
* Patients who undergo PPH technique along with another anorectal procedure.
* Patients with any other anorectal conditions, including fistula, anal fissure, inflammatory bowel disease, chronic diarrhea, or malignant lesions.
* Patients diagnosed with mucohemorrhoidal disease and experiencing acute complications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Postoperative improvement of symptoms of defecatory obstruction | 1 month
  Change From Baseline in Altomare Score and Agachan Wexner Score [Time Frame: 1 month]. Altomare Score: Assessed using an interviewer-led questionnaire with eight items (time spent at toilet, attempts to defecate each day, digitation, laxatives, enemas, straining, consistency, completeness), each rated on a 3- or 4-point Likert scale. Scores range from 0 (no symptoms) to 3 or 4 (severe symptoms), with a max score of 31 indicating obstructive defecatory syndrome (>3). Higher scores denote worse symptoms. Agachan Wexner Score: Derived from eight variables (Frequency of bowel movements, effort, Completeness, pain, time, assistance, failure, history), scored from 0 to 4 (except "assistance for defecation," 0-2). Global score is the sum, with >12 indicating constipation symptoms. Higher scores indicate worse defecatory obstruction symptoms.

SECONDARY OUTCOMES:
Postoperative change of the balloon expulsion test | 1 month
  Time recorded (<1 or >1 min) in ballon expulsion test in control and experimental group.
Postoperative change of the colonic transit time | 1 month
  Over 80% expulsion of 24 radiopaque markers on standing abdominal radiographs within five days

CONTACTS AND LOCATIONS:
Overall Officials: Cristopher Varela, MD, Principal Investigator — Instituto Venezolano de los Seguros Sociales
Locations (1):
- Hospital Domingo Luciani, Caracas, Miranda, Venezuela

IPD SHARING:
Plan to Share IPD: No